CLINICAL TRIAL: NCT05509556
Title: Effect Talocalcaneal Angle in Calcaneal Spur Formation
Brief Title: Talocalcaneal Angle in Calcaneal Spur Formation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021/141
Record Dates: First submitted 2022-08-08; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Foot Callus; Plantar Fascitis
Keywords: heel pain; talocalcaneal angle; calcaneal spur
MeSH Terms: conditions — Heel Spur

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with calcaneal spur on the lateral radiograph of the foot: The group in which talocalcaneal angle measurement was performed in patients with calcaneal spurs on the lateral radiograph of the foot.
  Interventions: Other: talocalcaneal angle measurement
- patients without calcaneal spur on lateral radiograph of the foot: The group in which talocalcaneal angle measurement was performed in patients without calcaneal spur on the lateral radiograph of the foot.
  Interventions: Other: talocalcaneal angle measurement

INTERVENTIONS:
Other: talocalcaneal angle measurement — talocalcaneal angle measurement on lateral foot radiographs

SUMMARY:
Calcaneal spur is one of the most common causes of chronic heel lower face pain without a traumatic cause. Obesity, sedentary life and advanced age play a role in its etiology. Mechanical overload is the main factor in the development of the disease. Impaired biomechanical factors in the foot cause repetitive microtraumas, traction periostitis and degenerative changes in the plantar fascia. The calcaneal spur is a result of this pathological process that creates pain. Many static radiological evaluation methods are used to evaluate the effect of foot anatomy in etiology. The talocalcaneal angle is one of them. It is the angle between the long axis of the talus and the long axis of the calcaneus. This angle shows the alignment of the back of the foot. It decreases with varus angulation of the back of the foot and increases with valgus angulation.

In this study, it was aimed to determine the place of the talocalcaneal angle values measured in the lateral radiographs of the foot in the etiology of painful calcaneal spur formation.

DETAILED DESCRIPTION:
The study was designed retrospectively. In this study, talocalcaneal angles of patients with heel pain and epin on lateral foot radiograph will be compared with talocalcaneal angle measurements on lateral foot radiographs without epin calcanei. Measurements will be made by the same physician, 3 measurements will be made and the average value will be recorded.

It was aimed to investigate the effect of talocalcaneal angle on calcaneal spur formation.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 30-75 who applied to our outpatient clinic with the complaint of pain with pressing on the heel for at least 3 months.

• Patients with calcaneal spur detected in the lateral radiographs of the feet

Exclusion Criteria:

Those who complain of heel pain for less than 3 months, have any rheumatological disease, have a previous history of foot and ankle fractures

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with lateral radiographs of the feet admitted to the hospital
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
talocalcaneal measurement on patient groups and control radiographs with heel spurs in the first | baseline
  On the lateral foot radiograph, the angle between the line drawn from the calcaneal tubercule to the 5th finger and the line drawn from the talus body to the calcaneal tubercule is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Aydeniz, 1, Principal Investigator — bakirkoy sadi konuk trainingandreseach hospital, Physical Therapy and rehabilitation department; Munevver Cinicioglu, Study Chair — bakirkoysadikonuk training and reseach hospital,Physical Therapy and rehabilitation department; Turker suleymanoglu, Study Chair — bakirkoysadikonuk training and reseach hospital,Physical Therapy and rehabilitation department; menekse gok, Study Chair — bakirkoysadikonuk training and reseach hospital,Physical Therapy and rehabilitation department; meltem vural, Study Chair — bakirkoysadikonuk training and reseach hospital,Physical Therapy and rehabilitation department
Locations (1):
- Bakirkorsadikonuk Training and Reseach Hospital, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No